CLINICAL TRIAL: NCT01470053
Title: A Multicenter, Randomized, Double-blind Phase Ⅲ Study of Mometasone Furoate/Azelastine Hydrochloride Combination Group and Mometasone Furoate and Azelastine Hydrochloride Group 4 Weeks After Treatment, Each Treatment Group Comparisons for Evaluation of Efficacy and Safety in Perennial Allergic Rhinitis Patient.
Brief Title: Efficacy and Safety of Mometasone Furoate Plus Azelastine HCl Combination Versus Mometasone Furoate Alone or Azelastine Alone in Patients With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL_NSFX_301
Record Dates: First submitted 2011-11-08; First posted 2011-11-11 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2011-11

CONDITIONS: Perennial Allergic Rhinitis
Keywords: mometasone furoate; azelastine HCl; perennial allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate; azelastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- mometasone furoate + azelastin HCl (Experimental): opaque suspension, four times each naris per day
  Interventions: Drug: mometasone furoate plus azelastine HCl
- mometasone furoate (Active Comparator): opaque suspension, four times each naris per day
  Interventions: Drug: mometasone furoate
- azelastine HCl (Active Comparator): lucidus colorless liquid, two times each naris per day
  Interventions: Drug: azelastine HCl

INTERVENTIONS:
Drug: mometasone furoate plus azelastine HCl
  Other Names: Nasaflex Nasal Spray
  Arms: mometasone furoate + azelastin HCl
Drug: mometasone furoate
  Other Names: NASONEX NASAL SPRAY
  Arms: mometasone furoate
Drug: azelastine HCl
  Other Names: AZEPTIN NASAL
  Arms: azelastine HCl

SUMMARY:
The purpose of this study is to evaluate of efficacy and safety of mometasone furoate plus azelastine HCl in patients with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 12 years of age
* Medical history of perennial allergic rhinitis for at least two years
* Moderate ro severe nasal symptom (during placebo run-in period AM rTNSS or PM rTNSS≥8)
* Positive skin prick test result within the previous 12 months

Exclusion Criteria:

* patients with active asthma that required therapy with inhaled or oral corticosteroids or long-term β-agonist
* patients with severe rhinostenosis, severely deviated nasal septum or local infection on the nasal mucous membrane
* patients with herpes zoster, glaucoma or cataract
* patients with history of operation or damage on nasal cavity or ocular region
* patients with drug-induced rhinitis
* patients with history of respiratory infection which requires antibiotic therapy within the previous 14 days
* Patients with lung disease including COPD
* Patients with history of immunotherapy or ongoing immunotherapy
* patients administered with super potent or potent corticosteroid
* patients administered with intra-muscular or intra-articular steroid within the previous 3 months
* patients administered with subcutaneous omalizumab within the previous 5 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
change from baseline in rTNSS(reflective Total Nasal Symptom Score) | 4 weeks

SECONDARY OUTCOMES:
change from baseline in AM rTNSS(AM reflective Total Nasal Symptom Score) | 4 weeks
change from baseline in PM rTNSS(PM reflective Total Nasal Symptom Score) | 4 weeks
change from baseline in iTNSS(instantaneous Total Nasal Symptom Score) | 4 weeks
change from baseline in AM iTNSS(AM instantaneous Total Nasal Symptom Score) | 4 weeks
change from baseline in PM iTNSS(PM instantaneous Total Nasal Symptom Score) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yang Gi Min, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea